CLINICAL TRIAL: NCT05291884
Title: Use of the Impella BTR™ in Patients With Heart Failure: An Early Feasibility Study
Acronym: BTR EFS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ABMD-CIP-21-01
Record Dates: First submitted 2022-02-11; First posted 2022-03-23 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Acute Decompensated Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Subjects receiving the Impella BTR (Experimental)
  Interventions: Device: Impella BTR

INTERVENTIONS:
Device: Impella BTR — Subjects will be prepared for pump insertion procedure according to clinical site standard of care. Procedural preparations for insertion of the Impella BTR are identical to the insertion of the Impella 5.0/5.5 via the axillary artery. The Impella BTR remains in situ until the patient is sufficiently recovered for removal or is transitioned to another form of support. It is expected that the Impella BTR is in situ for a maximum of 28 days.

SUMMARY:
This is a prospective, multi-center, single-arm, early feasibility study that aims to evaluate the safety of the Impella BTR™ in adult patients requiring left-ventricular hemodynamic support, and to evaluate the effectiveness of the Impella BTR™ in supporting patients to recovery or their next therapy.

DETAILED DESCRIPTION:
The objectives of this Early Feasibility Study are to evaluate the safety of the Impella BTR™ in adult patients requiring left-ventricular hemodynamic support. Additionally, to evaluate the feasibility of the Impella BTR™ in supporting patients to recovery or their next therapy. The investigational device consists of the following primary device and accessories: The Impella BTR™ Pump System (an intravascular transvalvular, micro-axial blood pump) and the Modified Automated Impella Controller™ (AIC) to allow control of the Impella BTR.

Following informed consent, subjects that meet all of the inclusion and none of the exclusion criteria, and in whom the Impella BTR™ is implanted or attempted to be implanted, will be considered enrolled into the Study. The device is inserted during a surgical procedure through a vascular graft that has been sutured onto the left or right axillary artery. After proper placement and passage through the aortic valve with the help of a guidewire, the device pumps blood from the left ventricle into the aorta. Once hemodynamic support is no longer required, the device is weaned and removed. Subjects will be followed to 90 days post-implant.

The primary and secondary endpoints will be summarized and presented without formal statistical testing. All adverse events including all Protocol-defined events, serious and non-serious, will be documented and reported from the time of subject enrollment until Study completion. Feasibility is defined as the ability of the pump to provide clinically adequate support for the duration of the implant up to 28 days. Clinically adequate support is defined as operating without device malfunctions or failures that result in device removal, replacement or use of an additional MCS device.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Subject has signed the Informed Consent
3. Subject has pre-existing heart failure, with NYHA Class IV prior to the index admission
4. Subject is presenting with acute heart failure and meets one of the following criteria:

   1. Sustained episode of systolic blood pressure ≤90 mmHg for at least 30 minutes or need for vasoactive agents to maintain such blood pressure
   2. Or a cardiac index (CI) <2.2 L/min/m2 determined to be secondary to cardiac dysfunction, in the absence of hypovolemia
   3. Or required support with an intra-aortic balloon pump

Exclusion Criteria:

1. Structural aortic valve regurgitation or stenosis of any grade greater than mild, with evidence of aortic sclerosis on pre-procedure echocardiography
2. New diagnosis of heart failure ≤90 days prior to enrollment
3. Previous aortic valve replacement or reconstruction
4. Prealbumin <150 mg/L (15 mg/dL) or Albumin <30 g/L (3 g/dL)
5. Thrombus in the left atrium or ventricle
6. STEMI ≤30 days prior to enrollment
7. Severe Cardiogenic Shock during index hospitalization - requiring multiple pressors, currently on mechanical circulatory support (not including IABP) or mechanical ventilation or experiencing PEA or refractory VT/VF
8. Unwitnessed cardiac arrest OR ≥30 minutes of CPR prior to enrollment OR any cardiac arrest with impairment in mental status, cognition or any global or functional neurological deficit.
9. Subjects with known aortic diseases
10. Any contraindication that precludes placing an Impella® including tortuous vascular anatomy, axillary artery diameter <7 mm
11. Infection of the proposed procedural access site or suspected systemic active infection
12. Known contraindication to heparin (i.e., heparin induced thrombocytopenia (HIT)), pork, pork products, contrast media or study required medication(s)
13. Intolerance to anticoagulant or antiplatelet therapies
14. History of bleeding diathesis or known coagulopathy, any recent GU or GI bleed or will refuse blood transfusions
15. Known hemoglobin diseases, such as sickle cell anemia or thalassemia
16. Subject is currently on dialysis
17. History of heart transplant
18. Prior cardiac surgery ≤90 days prior to enrollment
19. RV dysfunction requiring mechanical or inotropic support pre-device implant
20. History of stroke or intracranial hemorrhage ≤90 days prior to enrollment, or a history of cerebrovascular disease with significant (> 80%) uncorrected carotid stenosis, or any permanent neurological deficit
21. Restrictive or obstructive cardiomyopathy, constrictive pericarditis, restrictive pericarditis, pericardial tamponade
22. Pre-existing liver dysfunction defined as: Child-Pugh Class B or C
23. Pre-existing pulmonary disease requiring home oxygen
24. Suspected or known pregnancy
25. Subject has previously been symptomatic with or hospitalized for COVID-19 unless he/she has been discharged (if hospitalized) and asymptomatic for ≥8 weeks and has returned to his/her prior baseline (pre-COVID) clinical condition
26. Subject has other medical, social or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to give written informed consent and/or to comply with study procedures
27. Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device which has not reached its primary endpoint
28. Subject belongs to a vulnerable population [Vulnerable subject populations are defined as individuals with mental disability, persons in nursing homes, children, impoverished persons, homeless persons, nomads, refugees and those permanently incapable of giving informed consent.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility: successful hemodynamic support | Device explant or 28 days, whichever is shorter
  The ability of the pump to provide clinically adequate support for the duration of the implant up to 28 days. Clinically adequate support is defined as operating without device malfunctions or failures that result in device removal, replacement or use of an additional MCS device.
Safety: Major Device-Related Adverse Events | From date of enrollment to 28 days or discharge from hospital
  The rate of composite Major Device-Related Adverse Events

SECONDARY OUTCOMES:
Number of participants with Major Hemolysis | From date of enrollment to 28 days or discharge from hospital
All-cause mortality | From date of enrollment to 28 days or discharge from hospital & 90 days post-implant
Stroke | From date of enrollment to 28 days or discharge from hospital
Device malfunction | Device removal or up to 28 days
  That results in clinically inadequate support, not requiring removal, replacement or an additional device
Pump thrombus | Device removal or up to 28 days
Length of hospital stay | From date of enrollment to 28 days or discharge from hospital
Assessment of quality of life over baseline | Baseline to 90 days post-implant
  As measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ)

CONTACTS AND LOCATIONS:
Overall Officials: David D'Alessandro, MD, Principal Investigator — Massachusetts General Hospital; Jane Wilcox, MD MSc, Principal Investigator — Northwestern University Hospital
Locations (6):
- United States (6):
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cleveland Clinic, Cleveland, Ohio